CLINICAL TRIAL: NCT03437668
Title: Adjunctive Withania Somnifera (Ashwagandha) for Persistent Symptoms in People With Schizophrenia
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Unable to reach enrollment target due to COVID
Sponsor: Chengappa, K.N. Roy, MD (Other)
Collaborators: Stanley Medical Research Institute (Other); University of Maryland (Other)
Responsible Party: Principal Investigator, Stephen Marder, Professor, University of California, Los Angeles
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO18030276
Record Dates: First submitted 2018-02-01; First posted 2018-02-19 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Withania Somnifera
MeSH Terms: conditions — Schizophrenia | interventions — Ashwagandha

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Withania Somnifera Extract (WSE) (Experimental): WSE 500 mg bid for 12 weeks
  Interventions: Drug: WSE
- Placebo tablets (Placebo Comparator): Placebo oral tablet bid for 12 weeks
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: WSE — WSE tablets
  Other Names: Withania somnifera extracts; Ashwagandha; Sensoril®
  Arms: Withania Somnifera Extract (WSE)
Drug: Placebo Oral Tablet — Placebo tablet
  Arms: Placebo tablets

SUMMARY:
To determine whether a standardized extract of Withania somnifera will reduce psychopathology scores (PANSS total score) in persons with schizophrenia. A secondary aim is to determine whether WSE reduces measures of positive and negative symptoms (PANSS subscales) and stress scores on the Perceived Stress Scale (PSS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual (DSM) 5 diagnosis of schizophrenia or schizoaffective disorder
* Ability to provide informed written consent
* PANSS total score ≥ 70 or a CGI Severity Scored ≥ 4; and at least 2 positive symptom subscale items (i.e., delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, hostility and unusual thought content) scoring ≥ 4, or one of these items scoring ≥ 5, on a scale ranging from 1 = absent to 7 = extreme.
* Evidence of a positive symptom exacerbation during the year prior to study entry.
* For women of child bearing age, a negative serum pregnancy test at screening

Exclusion Criteria:

* Testing positive for illicit substances (positivity to marijuana or opioids will be assessed on a case by case basis due to the long elimination half life in the urine of marijuana and the use of opioids for various pain disorders, caffeine and nicotine are excepted)
* Receiving pharmacological treatment for addictions (naltrexone, suboxone, acamprosate, others) will be reviewed on a case by case basis
* Seriously unstable medical illnesses
* Pregnant or breast feeding women
* Known allergy or history of serious adverse event with WSE
* Subjects who may require imminent hospitalization (examples: suicidal or aggressive behavior)
* Currently receiving antibiotics, anti-viral, or anti-parasitic medications
* Currently receiving immunosuppressive medications (e.g. oral scheduled corticosteroids, chemotherapy or transplantation or HIV/AIDS associated drugs).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 47 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Marder, MD, Study Chair — Semel Inst at UCLA
Locations (2):
- United States (2):
  - UCLA, Los Angeles, California
  - Maryland Psychiatric Research Center, Catonsville, Maryland

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified will be submitted an NIH repository

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Withania Somnifera Extract (WSE) | Placebo Tablets
Started | 24 | 23
Completed | 20 | 19
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Withania Somnifera Extract (WSE) | Placebo Tablets | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (10.9) | 43.8 (12.1) | 43.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 18 | 20 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 22 | 21 | 43
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 9 | 14
  White | 16 | 12 | 28
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Symptom Scale
Description: The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of patients with schizophrenia. To assess a patient using PANSS, an approximately 45-minute clinical interview is conducted. The patient is rated from 1 to 7 on 30 different symptoms based on the interview as well as reports of family members or primary care hospital workers. Subjects can not score lower than 30 or higher than 210. Higher score indicates higher amount of psychopathology
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Withania Somnifera Extract (WSE) | Placebo Tablets
Number analyzed (Participants) | 22 | 21
score on a scale
  Week 0 | 65.0 (2.6) | 75.1 (2.6)
  Week 6 | 63.2 (2.4) | 72.0 (2.5)
  Week 12 | 61.3 (2.7) | 68.8 (2.7)
Statistical Analysis 1: Comparison: Withania Somnifera Extract (WSE) vs Placebo Tablets; Test type: Superiority — To test for a differential treatment effect, we fit a linear mixed with group, time, and a group by time interaction as the predictors and random intercepts to account for the correlations induced by the repeated measurements within subjects. Given the form of the trajectories and the small sample size, we chose to treat time as continuous to minimize the number of degrees of freedom and the risk of overfitting; p = .31, Mixed Models Analysis — p-value is for the interaction of time and treatment group in the mixed model; Slope = -0.22

2. Secondary Outcome: PANSS Negative Factor Score Also Know as Marder Factors
Description: The Marder negative factor is a factor-analysis derived dimension of the Positive and Negative Syndrome Scale (PANSS) that measures negative symptoms of schizophrenia. It's made up of seven items from the PANSS, including: Blunted affect, Emotional withdrawal, Poor rapport, Passive/apathetic withdrawal, Motor retardation, Active social avoidance, Lack of spontaneity in conversation. Each item is scored from 1 to 7 with a higher score indicating greater severity. Minimum score is 7 and maximum is 49
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Withania Somnifera Extract (WSE) | Placebo Tablets
Number analyzed (Participants) | 23 | 23
score on a scale
  Baseline | 2.05 (.84) | 2.68 (.67)
  12 weeks | 2.10 (.80) | 2.45 (.69)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Definitions consistent with clinicaltrials.gov
Arm/Group | Withania Somnifera Extract (WSE) | Placebo Tablets
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/24 | 3/23
Other Adverse Events (participants affected / at risk) | 12/24 | 18/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Withania Somnifera Extract (WSE) (N=24) | Placebo Tablets (N=23)
COVID 19 (Infections and infestations) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Withania Somnifera Extract (WSE) (N=24) | Placebo Tablets (N=23)
Objective tinnitus (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acid reflux (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Endometritis (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Back injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Weight loss (Investigations) | 1 (1) | 0 (0)
Decrease appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Auditory hallucinations (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT03437668/Prot_SAP_002.pdf